CLINICAL TRIAL: NCT00504491
Title: Rescue Treatment With Rituximab-CHOP Therapy and Alemtuzumab (R-CHOP-A) in Refractory or Recidivant Patients With Chronic Lymphocytic Leukemia After Purine-analogous Treatment
Brief Title: R-CHOP and Alemtuzumab in Patients With Chronic Lymphocytic Leukemia
Acronym: R-CHOP
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: IMP new owner decision
Sponsor: CABYC (Industry)
Collaborators: Francesc Bosch, MD (Unknown); Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other); Fundacion Clinic per a la Recerca Biomédica (Other); Bayer (Industry); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GELLC-2; 2007-003097-26 (EudraCT Number)
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Lymphocytic Leukaemia; Patients Resistant to a Purine Analogous; Patients Relapsed With Purines Therapy
Keywords: Rituximab-CHOP; Alemtuzumab; Chronic lymphocytic leukaemia
MeSH Terms: conditions — Leukemia, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Four Rituximab - CHOP courses will be given The courses will be given every 21 days Drug Dose Day Rituximab (Mabthera) 500mg/m2 1(*) (**) Cyclophosphamide 750mg/m2 1 Adriamycin 50mg/m2 1 Vincristine 1,4 mg/m2 1 Prednisone 60mg/m2 1 to 5
  (**) 1st course, 375 mg/m2 (*) If lymphocyte count is > 30 X 10 9/l, dose will be split up in two, which will be given in days 0 and 1
  Interventions: Drug: Rituximab-CHOP-Alemtuzumab

INTERVENTIONS:
Drug: Rituximab-CHOP-Alemtuzumab — Four Rituximab - CHOP courses will be given The courses will be given every 21 days

SUMMARY:
Since there is no standard rescue therapy for refractory CLL or relapsed to the purine analogous, our target is to carry out a rescue therapy combining several chemotherapy agents (CHOP) adding the synergistic effect of Rituximab in order to act against tumour-like CLL forms, with assessable size lymph nodes. Afterwards, based in other studies, we shall study the role of Alemtuzumab as drug for consolidation or improvement of responses obtained with the initial therapy (CHOP-R), acting by "cleaning" from peripheral blood and bone marrow the CLL lymphocytes that may have had remain as residual after chemotherapy induction therapy. More precisely, the addition of Alemtuzumab as maintenance treatment would increase the complete responses with negative residual disease number and may prolong the duration of the response. For this, it is necessary to have not only an adequate and rigorous clinical follow-up but also biological, i.e. being able to analyze minimal residual disease by molecular biology techniques. This is the reason of writing this phase II clinical trial protocol.

DETAILED DESCRIPTION:
OBJECTIVES

The objectives of this clinical trial are the following:

* Main objective of the study: Overall response rate obtained after R-CHOP regime followed by Alemtuzumab consolidation as second line therapy
* Secondary objectives

  * Determine the molecular complete response rate after R-CHOP regimen
  * Determine the efficacy of Alemtuzumab in response improvement after R-CHOP regimen: conversion of PR to CR and of MRD+ to MRD-.
  * Applicability (toxicity profile) of Alemtuzumab consolidation therapy.
  * As additional objectives will be considered:

    1. Prognostic value of several biological variables (ZAP-70 and cytogenetics) having influence on the response
    2. Response duration
    3. Progression free survival
    4. Overall survival

ELIGIBILITY:
Inclusion Criteria:

1. Patient's written informed consent before initiation of any specific procedure related with the study.
2. Age ≥ 18 years and ≤ 70 years
3. (ECOG) ≤ 2
4. Patients suffering from chronic lymphocyte leukaemia according to the established diagnostic criteria (Addendum A).
5. Active CLL defined by the presence of one or more of the following criteria:

   * Related symptoms: weight loss >10% in the 6 previous months, or fever >38ºC for 2 weeks with no evidence of infections, or extreme fatigue, or night sweats with no evidence of infection.
   * 5.2.Enlarged lymph nodes or giant node clusters (>10 cm in diameter) or progressive growth lymph nodes.
   * 5.3.Giant splenomegaly (> 6 cm under ribs border) or progressive splenomegaly.
   * 5.4.Progressive lymphocytosis (>50% increase in a period of 2 months) or lymphocyte duplication time (expected) < 6 months
   * 5.5.Proof of progressive bone marrow failure evidenced by development or worsening of anaemia and/or thrombopenia.
6. Patients previously treated in first line with purine analogous and showing:

   * Treatment failure (stable disease or progression)
   * Relapse within three years of therapy.
7. Agreement to use a high efficacy contraception method throughout all study period.

Exclusion Criteria:

1. Age > 70 years
2. Patients having received more than one therapy line
3. Patients that had not received previously purine analogous therapy.
4. CLL patients in transformation to more aggressive cytologic or pathologic forms (Pro-lymphocytic leukaemia large cell lymphoma, Hodgkin's lymphoma)
5. Hypersensitivity shown as anaphylactic reaction to any of the DRUGS used in the trial.
6. Patients with severe heart, lung, neurological, psychiatric or metabolic diseases not due to CLL
7. Patients under systemic and continued steroid therapy.
8. Impairment of renal function (Creatinine > 2 times the upper limit of normal) non-attributable to CLL.
9. Patients suffering anaemia or thrombocytopenia of autoimmune origin as well as those with a positive Coombs test
10. Impairment of liver function (Bilirubin, ASAT/ALAT or Gamma-GT > 2 times upper limit of normal) non attributable to CLL
11. Patients with active severe infectious disease
12. Patients suffering another malignancy (with the exception of focalized skin carcinoma)
13. Patients with positive serum tests for HBsAg or CHV
14. Patients with history of HIV or other severe immune depression conditions.
15. Pregnant or breast feeding women
16. Patients unable to attend the controls under outpatient regimen
17. Patients previously treated with alemtuzumab

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2012-01 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Response rate obtained after R-CHOP regimen followed by consolidation therapy with Alemtuzumab, as second line therapy. Haematological and non haematological toxicity will be graded in accordance with the WHO system | 57 months

CONTACTS AND LOCATIONS:
Overall Officials: Francesc Bosch, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (32):
- Spain (32):
  - Hospital de Son Dureta, Palma de Mallorca, Balearic Islands
  - ICO Badalona, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Valle de Hebron, Barcelona, Barcelona
  - ICO Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Althaia, Manresa, Barcelona
  - Corporacion Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital de Basurto, Bilbao, Bilbao
  - Hospital Marques de Valdecilla, Santander, Cantabria
  - Hospital Clinic i Provincial., Barcelona, Catalonia
  - ICO Gerona, Girona, Girona
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Gran Canaria
  - Hospital Virgen de las Nieves, Granada, Granada
  - Hospital Arnau de Vilanova, Lleida, Lleida
  - Hospital La Princesa, Madrid, Madrid
  - Hospital Gregorio Marañon, Madrid, Madrid
  - M.D.Anderson Internacional, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital 12 de octubre, Madrid, Madrid
  - Hospital Morales Meseguer, Murcia, Murcia
  - Hospital Clinico de Salamanca, Salamanca, Salamanca
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, Santiago de Compostela
  - Hospital Virgen del Rocio, Seville, Sevilla
  - Hospital Joan XXIII, Tarragona, Tarragona
  - Hospital Francisco de Borja, Gandia, Valencia
  - Hospital La Fe, Valencia, Valencia
  - Hospital Clinico de Valencia, Valencia, Valencia
  - Hospital Doctor Peset, Valencia, Valencia
  - Hospital General de Valencia, Valencia, Valencia
  - Hospital Miguel Servet, Zaragoza, Zaragoza